CLINICAL TRIAL: NCT04358991
Title: Pharmacokinetics of Ceftazidime-avibactam Among Critically-ill Patients Receiving Continuous Venovenous Hemodiafiltration
Brief Title: Pharmacokinetics of Ceftazidime-avibactam Among Critically-ill Patients Receiving CVVHDF
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Ryan Shields, Associate Professor, University of Pittsburgh
Other Study IDs: I# 0058410
Record Dates: First submitted 2020-04-17; First posted 2020-04-24 (Actual); Results first posted 2020-05-15 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — avibactam, ceftazidime drug combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples will be collected immediately before, and then at the following times thereafter intravenous administration of ceftazidime-avibactam: 1, 2, 4, 6, and 8 hours
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- invasive bacterial infections: patients who are receiving Ceftazidime-avibactam are asked to provide blood samples around a dosing of the medication for analysis of samples
  Interventions: Drug: Ceftazidime-avibactam

INTERVENTIONS:
Drug: Ceftazidime-avibactam — collection of blood samples around clinical dosing immediately pre-dose, then at the following times thereafter: 1, 2, 4, 6, 8, and 12 hours and EMR review.

SUMMARY:
Ceftazidime-avibactam is used for treatment of invasive Gram-negative bacterial infections among critically ill patients, including those on continuous venovenous hemodiafiltration . However, dosing of ceftazidime-avibactam for these patients remains undefined. The purpose of this study was to evaluate the pharmacokinetics of ceftazidime and avibactam among critically-ill patients, including those receiving CVVHD. This is a registration of Dr. Shields' exempt project under IRB approved research study STUDY19040363

DETAILED DESCRIPTION:
Patients who received ceftazidime-avibactam as part of their clinical care were consented. EMR data was collected as well as PK sampling around their dosing to include the following samples immediately pre-dose, then at the following times thereafter: 1, 2, 4, 6, and 8 hours. Blood samples were collected in lithium-heparin tubes from a central venous catheter that is not being used for the continuous venovenous hemodiafiltration. The tubes were centrifuged at 2500 rpm for 10 minutes within 1 hour from collection and the samples will be frozen at 80°C. The total concentrations of ceftazidime and avibactam were determined simultaneously from plasma by using a validated HPLC-tandem MS assay. Noncompartmental pharmacokinetics were calculated using the linear-up and logarithmic-down trapezoidal method, based on the assumption of first-order elimination.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients receiving ceftazidime-avibactam as standard care

Exclusion Criteria:

* Less than 18 years-old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with confirmed or presumed invasive bacterial infections
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Shields, Pharm D, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared through peer-reviewed publication
Supporting Information: CSR
Time Frame: Within 1 year of study completion
Access Criteria: will be on clinicaltrials.gov

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Included: 20 patients meeting inclusion criteria were enrolled into the trial
Period: Overall Study
Arm/Group | Subjects Included
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Included
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Serum Levels of Ceftazidime and Avibactam Among Critically-ill Patients
Description: PK samples obtained around standard of care dosing regimens immediately before and at 1, 2, 4, 6, and 8 hours after administration
Time Frame: 8 hours
Measure: Median (Inter-Quartile Range); unit: mcg/mL
Arm/Group | Subjects Included
Number analyzed (Participants) | 20
mcg/mL
  Ceftazidime Cmax | 80.6 [61.2 to 104.1]
  Avibactam Cmax | 15.9 [11.8 to 23.0]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored until the end of ceftazidime-avibactam treatment, up to 14 days
Arm/Group | Subjects Included
All-Cause Mortality (participants affected / at risk) | 3/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT04358991/Prot_SAP_000.pdf